CLINICAL TRIAL: NCT03536624
Title: Effects of a Thermal Spa Short Residential Program for Prevention of Work-related Stress / Burn-out on Biomarkers of Stress - A Proof of Concept Study
Acronym: ThermStress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Regional Council of Auvergne-Rhône-Alpes (Other); European Regional Development Fund (Other); Spa resort of Néris-les-Bains, SEMETT, 6 place des Thermes, 03310 Néris-les-Bains, France (Unknown); Université d'Auvergne (Other); LaPEC laboratory (EA 4278), Avignon University, Avignon, France (Unknown); Innovatherm (Industry); EIPAS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHU-386; 2016 A02082 49 (Other: 2016 A02082 49)
Record Dates: First submitted 2018-03-26; First posted 2018-05-24 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Stress; Burn Out; Heart Rate Variability
Keywords: prevention; biomarkers; stress; burn out; occupation; work; spa bath
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Masking Description: no masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Participants will be involved in a short-term spa residential program of 6 days combining psychological intervention, physical activity, thermal spa treatment, health education and corrections of eating disorders.
  After the program, participants will be followed for 12 months.
  Interventions: Behavioral: 6 days spa residential program

INTERVENTIONS:
Behavioral: 6 days spa residential program — 6 days spa residential program combining psychological intervention, physical activity, thermal spa treatment, health education and corrections of eating disorders.

SUMMARY:
Work-related stress is a public health issue. Among the multiple physical and psychological consequences of stress, increased mortality and cardiovascular morbidity seem the main concern. The thermal spa resort of Néris-Les-Bains is one of the five spa resorts in France specialized in the treatment of psychosomatic disorders. Among all these resorts proposing a thermal residential program of three weeks, only one thermal spa resort (Saujon) has a program for occupational burn-out. However, a shorter thermal spa residential program seems more compatible with professional context (availability of individuals), and focusing on work-related stress prevention (before the state of burn-out).

The main hypothesis is that a short thermal spa residential program (6 days) of work-related stress prevention will exhibit its efficacy through objective measures of well-being and cardiovascular morbidity.

DETAILED DESCRIPTION:
The Therm-Stress protocol was designed to provide a better understanding of the effect of a short spa residential program of work-related stress prevention on the improvement of heart rate variability.

In the present protocol, parameters are measured on six occasions (inclusion, 6 days before the start, at the start of the spa, at the end of the spa, at 6 months and at 12 months).

Statistical analysis will be performed using Stata software (version 13; Stata-Corp, College Station, Tex., USA). All statistical tests will be two-sided and p<0.05 will be considered significant. After testing for normal distribution (Shapiro-Wilk test), data will be treated either by parametric or non-parametric analyses according to statistical assumptions. Inter-groups comparisons will systematically be performed 1) without adjustment and 2) adjusting on factors liable to be biased between groups.

Analysis will be performed using anova or Kruskal-Wallis (KW) tests. When appropriate (p<0.05), a post-hoc test for multiple comparisons (Tukey-Kramer after anova and Dunn post KW) will be used. Linear regression (with logarithmic transformation if necessary) considering an adjustment on covariates fixed according to epidemiological relevance and observance to physical activity will complete the analysis.

Comparisons of categorical variables will be performed using Chi-squared or Fischer test. Marascuillo's procedure will be performed for multiple comparisons. Relations between quantitative outcomes will be analyzed using correlation coefficients (Pearson or Spearman). Fisher's Z transformation and William's T2 statistic will be performed to compare correlations between variables and within a single group of subjects. Longitudinal data will be treated using mixt-model analyses in order to treat fixed effects group, time and group x time interaction taking into account between and within participant variability.

ELIGIBILITY:
Inclusion Criteria:

* Workers with a visual analog scale of stress greater than 50 mm
* from 18 years to retirement
* written informed consent
* Affiliation to French health care system (for France)

Exclusion Criteria:

* Participant refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
heart rate variability | at inclusion (Month1 to Month5)
  To assess the ability of a short spa residential program of management of work-related stress in increasing heart rate variability, a biomarker of both stress and morbidity/mortality.
  Heart rate variability will be measured by zephyr during 26h recording time

SECONDARY OUTCOMES:
Variation of biomarkers of stress after the end of the interventional phase. | at inclusion (Month1 to Month5)
  Evaluate the effectiveness of an individualized thermal intervention on biomarkers of stress among working people.
Variation of cardiovascular risk after the end of the interventional phase. | at inclusion (Month1 to Month5)
  Evaluate the effectiveness of an individualized thermal intervention on cardiovascular risk among working people.
Genetic polymorphisms related to stress | at inclusion (Month1 to Month5)
  effectiveness of an individualized thermal intervention on genetic polymorphisms related to stress.
Demographics information | at inclusion (Month1 to Month5)
  Demographics information will be obtained via a single questionnaire including questions on age, gender, qualification, personal work status, ethnicity, life and occupational events
Variation of health factors risks after the interventional phase | at inclusion (Month1 to Month5)
  Evaluate the effectiveness of an individualized thermal intervention on health factors.
Variation of body composition after the interventional phase | at inclusion (Month1 to Month5)
  Evaluate the effectiveness of an individualized thermal intervention on body composition.
Variation of subjective stress measures after the interventional phase | at inclusion (Month1 to Month5)
  Evaluate the effectiveness of an individualized thermal intervention on subjective stress measures.
Variation of health biomarkers after the interventional phase | at inclusion (Month1 to Month5)
  Evaluate the effectiveness of an individualized thermal intervention on Health-related risk assessed by biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic DUTHEIL, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France